CLINICAL TRIAL: NCT01204957
Title: Brown Seaweed as a Breast Cancer Preventive
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Principal Investigator, Jane Teas, Professor, University of South Carolina
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: USCIRB#060701
Record Dates: First submitted 2010-09-16; First posted 2010-09-17 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-04

CONDITIONS: Breast Cancer
Keywords: Homocysteine; Insulin-like growth factor; Insulin-like growth factor binding protein; Serum estrogen; Urinary phytoestrogens; Thyroid hormones
MeSH Terms: conditions — Breast Neoplasms | interventions — Soybean Proteins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 Seaweed and Soy Protein (Experimental): Arm 1 5 g/d Seaweed for 6 wk, then 5 g/d Seaweed and Soy Protein for 1 wk
  Interventions: Dietary Supplement: Seaweed and Soy Protein
- Arm 2 Placebo and soy protein (Experimental): Arm 2 5 g/d Placebo for 6 wk, then 5 g/d Placebo and Soy Protein for 1 wk
  Interventions: Dietary Supplement: Placebo and Soy Protein

INTERVENTIONS:
Dietary Supplement: Seaweed and Soy Protein — 5 g/d Seaweed for 6 wks, followed by 5 g/d Seaweed + Soy Protein for 1 wk
  Other Names: Solae Soy Food Ingredient Powder (AB1.2 HG 20CA 29); Alaria esculenta
  Arms: Arm 1 Seaweed and Soy Protein
Dietary Supplement: Placebo and Soy Protein — 5 g/d Placebo for 6 wks, followed by 5 g/d Placebo + Soy Protein for 1 wk
  Other Names: Solae Nutritious Food Ingredient Powder (AB1.2 HG 20CA 29); Maltrin M100 maltodextrin (Grain Processing)
  Arms: Arm 2 Placebo and soy protein

SUMMARY:
Japanese postmenopausal women in Japan have about one ninth the rate of American postmenopausal women. Rates of breast cancer double even after just ten years among Japanese women who migrate to the US. Diet is thought to be an important factor, and the investigators were interested in whether dietary seaweed, with and without soy supplements, could influence known biomarkers of breast cancer risk in American women.

DETAILED DESCRIPTION:
33 healthy postmenopausal women were randomized to 6 wk seaweed then 1 wk seaweed plus soy or 6 wk placebo then 1 wk placebo plus soy. Blood and urine samples were collected at the end of each treatment period and analyzed for estrogen, homocysteine, antioxidants, insulin-like growth factors and thyroid hormones. Urine was analyzed for phytoestrogens and iodine.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal (self-reported cessation of menstruation 1 y prior to enrollment)
* If breast cancer survivor, all therapy completed at least 6 months prior to enrollment
* Agreed to eat their normal diet, avoiding seaweeds and phytoestrogen-rich foods,
* Restricting alcoholic intake to #2 drinks (24 g alcohol)/wk -Continuing habitual intake of vitamins, supplements, and medications during the study. -

Exclusion Criteria:

* No allergies to seaweed, soy, shellfish, or iodine
* No current use of tobacco;
* No thyroid dysfunction or treatment within the previous 5 y;
* Negative thyroid peroxidase antibodies as determined by screening;
* No hormone replacement therapy or for breast cancer survivors, no chemotherapy or radiation treatments within the preceding 6 mo
* No history of cancer (other than breast cancer)
* No current gastrointestinal disorders or diabetes; omnivorous eating habits, including meat and dairy products at least twice/wk
* No oral antibiotics, iodine containing medications, or corticosteroids treatment within the previous 3 mo.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 1998-10; Primary Completion 1999-03 (Actual); Study Completion 1999-03 (Actual)

PRIMARY OUTCOMES:
Thyroid hormones affected by dietary seaweed and soy supplements | 14 weeks
  6 wk seaweed followed by 1 wk seaweed plus soy; Or 6 wk placebo followed by 1 wk soy 3 wk washout period then crossover to alternate arm

SECONDARY OUTCOMES:
Serum estrogen and urinary phytoestrogen concentrations affected by seaweed and soy | 14 wks
  6 wk seaweed then 1 wk seaweed plus soy; OR 6 wk placebo then 1 wk soy 3 wk washout period, then crossover to alternate arm
Serum antioxidant and homocysteine concentrations associated with seaweed and soy | 14 wks
  6 wks seaweed followed by 1 wk seaweed plus soy OR 6 wk placebo followed by 1 wk soy 3 wk washout period, then crossover to alternate arm
Serum IGF-1 and IGFBP3 changes associated with seaweed and soy supplementation | 14 wk
  6 wk seaweed then 1 wk seaweed plus soy OR 6 wk placebo then 1 wk soy plus placebo 3 wk washout then crossover to alternate arm

CONTACTS AND LOCATIONS:
Overall Officials: Jane Teas, Ph.D., Study Director — University of South Carolina
Locations (1):
- University of Massachusetts, Worcester, Massachusetts, United States

REFERENCES:
- [Result] Teas J, Hurley TG, Hebert JR, Franke AA, Sepkovic DW, Kurzer MS. Dietary seaweed modifies estrogen and phytoestrogen metabolism in healthy postmenopausal women. J Nutr. 2009 May;139(5):939-44. doi: 10.3945/jn.108.100834. Epub 2009 Mar 25. PMID 19321575
- [Result] Teas J, Braverman LE, Kurzer MS, Pino S, Hurley TG, Hebert JR. Seaweed and soy: companion foods in Asian cuisine and their effects on thyroid function in American women. J Med Food. 2007 Mar;10(1):90-100. doi: 10.1089/jmf.2005.056. PMID 17472472
- [Result] Teas J, Pino S, Critchley A, Braverman LE. Variability of iodine content in common commercially available edible seaweeds. Thyroid. 2004 Oct;14(10):836-41. doi: 10.1089/thy.2004.14.836. PMID 15588380